CLINICAL TRIAL: NCT03914885
Title: Compassionate Use Re-Infusion of ATLCAR.CD30
Status: No longer available | Type: Expanded Access
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1907-ATL-COM
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2019-12

CONDITIONS: Hodgkin Lymphoma, Adult
MeSH Terms: conditions — Hodgkin Disease | interventions — Bendamustine Hydrochloride; fludarabine; fludarabine phosphate

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Genetic: ATLCAR.CD30 — Administered at a dose of 2 x 10^8 cells/m2
  Other Names: CD30 CAR T cells
Drug: Bendamustine — Administered as a dose of 70mg/m2/day over 3 consecutive days; maybe dose reduced per treating physician discretion based on prior toxicities and the patient's clinical status
  Other Names: Bendeka; Treanda
Drug: Fludarabine — Administered at a dose of 30mg/m2/day over 3 consecutive days; given concomitantly with bendamustine
  Other Names: Fludara

SUMMARY:
This protocol for compassionate use combines 2 different ways of fighting disease: antibodies and T cells. Both antibodies and T cells have been used to treat patients with cancers, and both have shown promise, but neither alone has been sufficient to cure most patients. This protocol combines both T cells and antibodies to create a more effective treatment. The investigational treatment is called autologous T lymphocyte chimeric antigen receptor cells targeted against the CD30 antigen (ATLCAR.CD30) administration.

Prior studies have shown that a new gene can be put into T cells and will increase their ability to recognize and kill cancer cells. The new gene that is put in the T cells in this study makes a piece of an antibody called anti-CD30. This antibody sticks to leukemia cells because they have a substance on the outside of the cells called CD30. For this protocol, the anti-CD30 antibody has been changed so that instead of floating free in the blood part of it is now joined to the T cells. When an antibody is joined to a T cell in this way it is called a chimeric receptor. These CD30 chimeric (combination) receptor-activated T cells seem to kill some of the tumor, but they do not last very long in the body and so their chances of fighting the cancer are unknown.

The primary purpose of this protocol is to treat a single patient with a second dose of ATLCAR.CD30 T cells.

DETAILED DESCRIPTION:
Lymphodepleting Chemotherapy:

The patient will receive a lymphodepleting regimen of bendamustine 70mg/m2/day over 3 consecutive days and fludarabine 30mg/m2/day over 2 consecutive days. Bendamustine and fludarabine will be administered concomitantly. Dose reduction of bendamustine may occur per treating physician discretion based on prior toxicities and the clinical status of the patient.

Administration of ATLCAR.CD30 T cells:

Post lymphodepletion, if the patient meets eligibility criteria for cellular therapy, then will receive ATLCAR.CD30 T cells within 2-14 days after completing the pre-conditioning chemotherapy regimen. We will administer ATLCAR.CD30 T cells post lymphodepletion at a dose of 2 x 10^8 cells/m2.

Duration of Therapy:

Therapy under this compassionate use protocol involves 1 infusion of ATLCAR.CD30 cells.

Duration of Follow-up:

The patient will be followed for up to 15 years for replication-competent retrovirus evaluation or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky or Lansky score of >60%.
* WOCBP must be willing to use 2 methods of birth control or be surgically sterile , or abstain from heterosexual activity for the course of the study, or for 6 months after the study is concluded. WOCBP are those who have not been surgically sterilized or have not been free from menses for > 1 year. The two birth control methods can be composed of: two barrier methods or a barrier method plus a hormonal method to prevent pregnancy. WOCBP subjects will also be instructed to tell their male partners to use a condom.
* Must not be pregnant or lactating.
* Must not have tumor in a location where enlargement could cause airway obstruction.
* Must not have current use of systemic corticosteroids at doses ≥10 mg prednisone daily or its equivalent; those receiving <10mg daily may be enrolled at discretion of the Investigator
* Evidence of adequate organ function as defined by:

  * ANC>1.0 × 109/L
  * Platelets >75 × 109/L
  * Total bilirubin ≤2 × ULN, unless attributed to Gilbert's syndrome
  * AST ≤3 × ULN
  * Serum creatinine ≤1.5 × ULN
  * Pulse oximetry of >90% on room air Note: Patient may receive a second infusion without prior lymphodepletion if they meet the eligibility criteria in this Sections 3.1 and 3.2 at the time of infusion, but do not meet the eligibility requirements for adequate bone marrow function and platelet counts
* Negative serum pregnancy test within 72 hours prior to lymphodepletion or documentation that the patient is post-menopausal. Post-menopausal status must be confirmed with documentation of absence of menses for > 1 year or documentation of surgical menopause involving bilateral oophorectomy.
* Patient cannot be on strong inhibitors of CYP1A2 (e.g., fluvoxamine, ciprofloxacin) as these may increase plasma concentrations of bendamustine, and decrease plasma concentrations of its metabolites. See http://medicine.iupui.edu/clinpharm/ddis/ for an updated list of strong inhibitors of CYP1A2. (This applies to subjects who receive bendamustine for lymphodepletion (required) up through 72 hours after the last dose of bendamustine)
* Patient is a good candidate for treatment with ATLCAR.CD30 per the investigator's discretion.

Exclusion Criteria:

* No evidence of uncontrolled infection or sepsis.
* Evidence of adequate organ function as defined by:

  * Total bilirubin ≤2 × ULN, unless attributed to Gilbert's syndrome
  * AST ≤3 × ULN
  * ALT ≤3 × ULN
  * Serum creatinine ≤1.5 × ULN
  * Pulse oximetry of >90% on room air
* Patient has no clinical indication of rapidly progressing disease in the opinion of the treating physician
* Patient is a good candidate for treatment with ATLCAR.CD30 per the investigator's discretion.
* If Patient has had positive hepatitis B core antibody testing while on the LCCC 1532-ATL clinical trial, they must not have had re-activation of the Hepatitis B virus since baseline testing (i.e., they will be excluded if any of their hepatitis B viral load testing is positive up until the point of eligibility determination for re-infusion).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Grover, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, North Carolina, United States